CLINICAL TRIAL: NCT02911727
Title: Fast-track Discharge After Elective Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herning Hospital (Other)
Responsible Party: Principal Investigator, Anne Kruse, MD, Herning Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1
Record Dates: First submitted 2016-09-02; First posted 2016-09-22 (Estimated); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Postoperative Period
Keywords: Cesarean section; Postnatal Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fast-track discharge (Experimental): Intention to discharge within 28 hours after elective cesarean section including a home visit by a nurse or midwife from the postnatal ward.
  Interventions: Procedure: Fast-track discharge
- Standard discharge (No Intervention): Discharge at least 48 hours after elective cesarean section.

INTERVENTIONS:
Procedure: Fast-track discharge — As described above
  Arms: Fast-track discharge

SUMMARY:
Cesarean section (CS) is a procedure with prolonged hospital stay compared to the routine for normal vaginal delivery in multiparas. The difference is caused mainly by postoperative pain but improvements in management of pain may change this situation and make early discharge possible. However, several aspects need to be considered.

The aim of this project is to evaluate fast-track discharge for multiparas after elective CS concerning neonatal and maternal complications as well as the parents' sense of security and well-being.

The study is a randomized controlled trial including 142 women allocated to either 1) the intention to discharge within 28 hours followed by a home visit or 2) standard discharge after at least 48 hours after elective CS.

This study will be among the first evaluating fast-track discharge after CS in a European context. If a positive outcome is achieved, we expect that fast-track discharge can be implemented with improved quality and reduced costs in postnatal care following elective CS.

ELIGIBILITY:
Inclusion Criteria:

* Planned elective CS of multiparous women
* Singleton pregnancy
* Gestational age at least 37+0 weeks
* Prepregnancy BMI <35

Exclusion Criteria:

* Lack of consent
* Women with no or little understanding of and ability to speak Danish
* Expected maternal or neonatal complications after delivery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2016-10; Primary Completion 2019-12-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Parents' Postnatal Sense of Security | Measured one week after delivery
  Using the validated PPSS-questionaire

SECONDARY OUTCOMES:
Pain scores | During the first week postpartum
  Measured by the patient in a questionnaire using numeric rating scale
Use of analgesia | During the first week postpartum
  Daily consumption in mg of paracetamol, NSAID and opioid.
Mobilization | 5 days postpartum
  Step count measured by an activity monitor (Fitbit Flex)
Breastfeeding | 6 months after delivery
  Duration and extent of breastfeeding
Readmissions | 28 days postpartum
  Number of readmissions and length of hospital stay in number of days
Surgical complications | 28 days postpartum
  Number of complications using the Clavien-Dindo Classification (1-5)
Complications in the postnatal period | 28 days postpartum
  Number and type of complications using the ICD-10 classification
Contacts to the health care system | 28 days postpartum
  Number of contacts and site of contacts (primary or secondary care)

CONTACTS AND LOCATIONS:
Overall Officials: Byrjalsen, MD, Study Chair — Department chairman
Locations (1):
- Department of Obstetrics and Gynecology, Herning, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jones E, Stewart F, Taylor B, Davis PG, Brown SJ. Early postnatal discharge from hospital for healthy mothers and term infants. Cochrane Database Syst Rev. 2021 Jun 8;6(6):CD002958. doi: 10.1002/14651858.CD002958.pub2. PMID 34100558